CLINICAL TRIAL: NCT04028037
Title: Clinical Comparison of Full-thickness Palatal Graft Technique (FTPGT) vs Coronally Advanced Flap With Subepithelial Connective Tissue Graft (CAF+SCTG)in Obtaining Complete Root Coverage: a Randomised Controlled Study
Brief Title: Effectiveness of Full-thickness Palatal Graft Technique (FTPGT) in Obtaining Complete Root Coverage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: G. d'Annunzio University (Other)
Responsible Party: Principal Investigator, Michele Paolantonio, Head of Periodontology, G. d'Annunzio University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: uchieti2
Record Dates: First submitted 2019-07-17; First posted 2019-07-22 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Custom made computer-generated table provides the randomly allocation of experimental unit in the two groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FTPGT treated patients (Experimental): The recipient site will be prepared according to Langer&Langer modified technique, raising a split-thickness flap without vertical incisions. The harvest of palatal graft will be done using FTPG technique ant it will be made up of an apico-lateral portion of connective tissue and periosteum, and of a full-thickness central "U" shaped part.The palatal graft will be adapted to the recipient site and sutured.
  Interventions: Procedure: FTPGT treated patients
- CAF+SCTG treated patients (Active Comparator): A tension-free trapezoidal flap will be elevated by the split-full-split technique. A 1-mm thick SCTG will be harvested from the palate as epithelialized graft. After epithelium removal, the graft was positioned and sutured 1mm apical to the cement-enamel junction with 5-0 resorbable sutures . The SCTG will then be covered by the tension-free coronally positioned flap by 5-0 silk sutures.
  Interventions: Procedure: CAF+SCTG treated patients

INTERVENTIONS:
Procedure: FTPGT treated patients — The recipient bed will be prepared according to Langer&Langer modified technique. Intrasulcular incision will be performed from at least one tooth mesial and one tooth distal to the tooth with gingival recession, without vertical incisions.A split-thickness flap will be raised.The harvest of palatal graft will be done using FTPG technique. An incision, parallel to the gingival margin, deep to the bone, will be made. At the center of this incision, a "U" shaped one about 1-2mm deep will made, with the convex side towards the palatine vault.The width of the "U" incision will be equal to the width of the GR and the length will be 1mm greater.A split-thickness dissection of the area surrounding the "U" shaped incision will be done.The graft will be removed by detaching it from the bony surface.The graft will be made up of an apico-lateral portion of connective tissue and periosteum, and of a full-thickness central part.The palatal graft will be adapted to the recipient site and sutured.
  Arms: FTPGT treated patients
Procedure: CAF+SCTG treated patients — According to De Sanctis & Zucchelli, a tension-free trapezoidal flap will be elevated by the split-full-split technique and the anatomic papillae will be de-epithelialized. A 1-mm thick SCTG will be harvested from the palate as epithelialized graft. The height of the graft was equal to the distance between the buccal bone crest and the CEJ. After epithelium removal, the graft was positioned and sutured 1mm apical to the cement-enamel junction with 5-0 resorbable sutures . The SCTG will then be covered by the tension-free coronally positioned flap, sutured about 2mm over the CEJ by 5-0 silk sutures.
  Arms: CAF+SCTG treated patients

SUMMARY:
In this randomized controlled clinical trial we will compare the clinical outcome of Full thickness palatal graft technique (FTPGT) to coronally advanced flap (CAF) + subepithelial connective tissue graft (SCTG) in the treatment of RT1 (Cairo et al. classification) recessions.

Forty patients, presenting at least one RT1 recession, will be treated with bilaminar procedures . 20 participants will receive FTPGT approach (test group) and 20 patients will undergo CAF+SCTG (control group). Complete root coverage (CRC) will be assumed as the main outcome at 12 months after treatment. Gingival recession (GR), clinical attachment level (CAL), pocket depth (PD), keratinized tissue width (KT,) thickness of keratinized tissue (GT) will be assessed at baseline and 12 months after treatment. Patient-reported outcome measures (PROMs) will be reported: namely, the number of painkiller tablets taken during the first week, the degree of general discomfort (D) experienced assessed on a VAS scale (0-10), the extent of changes in their eating habits (CFH), dentin hypersensitivity (DH), patient-reported aesthetic satisfaction (PRES) quantified on a VAS scale (0-10) and overall treatment satisfaction (OTS).

DETAILED DESCRIPTION:
This study will be a prospective, randomized and controlled clinical trial designed to compare two modalities of treatment of RT1 recessions: FTPG versus CAF+SCTG. From each patient study one RT1 recession will be included. Clinical parameters will be evaluated at baseline and 12 months after treatment.

40 patients seeking treatment at the Unit of Periodontology of the University of Chieti, Pescara, Italy, and affected by RT1 recessions will be selected for the study.

All 40 patient will undergo a professional supra-gingival scaling by ultrasonic instruments. To each patient motivational oral home care instructions in order to acquire correct and pressure-less brushing technique and a-traumatic use of dental floss and/or inter-dental brush will be given. In addition electric toothbrush use with controlled pressure with extra-soft head will be suggested and instructions about it will be conferred. Only the achievement of supra-gingival plaque control through a-traumatic oral hygiene procedures will permit the access of the surgical step.

Custom made computer-generated table provides the randomly allocation of experimental unit in the two groups.

The post-surgical care will be founded for all patients on 2 g/day amoxicillin plus clavulanic acid for 6 days, oral ketoprofen for pain-control if needed . Two weeks after surgery suture will be removed. Plaque control of grafted area will be performed for 3 weeks after surgery through a double rinse in a day with 0.12% chlorhexidine digluconate solution. Furthermore, the patients will use a 1% chlorhexidine gel twice daily. Patients underwent weekly supragingival hygiene and motivational reinforcement for 6 weeks. Cautious brushing by a soft toothbrush and interdental brushing will be recommended only 2 weeks after sutures removal.

All measurements will be performed by a single experienced operator. Complete root coverage (CRC) will be assumed as the main outcome at 12 months after treatment. Gingival recession (GR), clinical attachment level (CAL), pocket depth (PD), keratinized tissue width (KT,) thickness of keratinized tissue (GT) will be assessed at baseline and 12 months after treatment.

PROMs will also be evaluated. That is, patients will be asked to write down the number of painkiller tablets (400 mg of ibuprofen) taken during the study the first week.

The degree of general discomfort (D) experienced will be assessed on a VAS scale (0-10), and the extent of changes in their eating habits (CFH) caused by the palate will be indicated wound. Dentin hypersensitivity (DH) will be evaluated at T0 and T1 according to a scale from 0 to 3 (0" reaction to the air stimulus; "1" reaction without requiring its termination; "2" reaction and request to stop it; "3" painful stimulus complaint).

Patient-reported aesthetic satisfaction (PRES) at T1 will also be quantified on a VAS scale (0-10). Overall treatment satisfaction (OTS) at T1 will be assessed by asking each patient if they would undergo surgery again (yes/no).

ELIGIBILITY:
Inclusion Criteria:

* systemic factors (no systemic diseases; no coagulation disorders; no medications affecting periodontal status in the previous 6 months; no pregnancy or lactation
* never smokers/former smokers >=10years
* a full-mouth plaque score (FMPS)and a full-mouth bleeding score (FMBS) lower than 15%
* no periodontal surgery on the experimental sites
* >= 20 teeth without mobility
* no presence of cervical carious lesions or periapical lesions at experimental sites
* at leat one RT1 buccal gingival recession

Exclusion Criteria:

* systemic diseases
* coagulation disorders
* medications affecting periodontal status in the previous 6 months
* pregnancy or lactation
* Smokers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Percentage (%) of Complete Root Coverage (CRC) | 12 months
  Percentage of teeth with CRC determined with the following formula: T0 GR-T1 GR/T0 GR.

SECONDARY OUTCOMES:
Clinical Attachment Level (CAL) | 12 months
  Distance between cementoenamel junction(CEJ) and depth of the pocket
Pocket Depth (PD) | 12 months
  Distance between gingival margin and depth of the pocket
Gingival Thickness (GT) | 12 months
  Gingival thickness (GT) was measured 1 mm apical to the sulcus depth, perpendicular to the gingiva until bone, using an endodontic K-file. GT was the distance from the tip of the K-file to the silicon disk.
Keratinized Tissue width (KT) | 12 months
  Distance between gingival margin and mucogingival junction
Number of painkiller tables | First week after surgery
  Number of painkiller tablets taken during the first week.
Overall Discomfort (D) | 2 weeks after surgery
  Overall discomfort experienced, reported on a VAS scale (0-10)
Feeding Habits Changes (CFH) | 2 weeks after surgery
  Extent of the feeding habits changes (CFH) caused by the palatal wound.
Dentine hypersensitivity (DH) | 12 months
  Dentine hypersensitivity evaluated using Schiff cold air sensitivity scale
Patient-Reported Esthetic Satisfaction (PRES) | 12 months
  Patient-reported esthetic satisfaction (PRES) quantified on a VAS scale (0-10), will be recorded after observing simultaneously 2 standardized photographs showing the treated site +2 mesial and 2 distal teeth and the MGJ.
Overall Treatment Satisfaction (OTS) | 12 months
  Overall Treatment Satisfaction (OTS) will be assessed by asking each patient if he would undergo surgery again (yes/no).

CONTACTS AND LOCATIONS:
Overall Officials: michele paolantonio, Principal Investigator — università G. D'annunzio Chieti-Pescara
Locations (1):
- G. d'Annunzio University, Chieti, CH, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Paolantonio M, De Ninis P, Santamaria P, Balice G, Serroni M, Sinjari B, Frisone A, Di Gregorio S, Romano L, Murmura G, Femminella B. Clinical comparison of two surgical techniques in obtaining complete root coverage of single RT1 gingival recessions. Clin Oral Investig. 2025 Sep 10;29(10):444. doi: 10.1007/s00784-025-06491-2. PMID 40928531